CLINICAL TRIAL: NCT00928434
Title: A Randomized, Controlled, Open-Label Study Investigating the Safety and Efficacy of Degarelix Given Intermittently vs Continuous Androgen Deprivation Therapy With Lupron or Degarelix in Patients With Prostate Cancer With Prior Treatment Failure After Localized Treatment
Brief Title: A Study of Degarelix in Patients With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FE200486 CS37
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Results first posted 2016-12-13 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- DI (Degarelix Intermittent) (Experimental): Patients in this arm received degarelix with a starting dose of 240 mg at a concentration of 40 mg/mL on Day 0 administered subcutaneously (s.c.) into the anterior abdominal wall via two equivalent injections of 120 mg (3 mL) each.
  Six maintenance doses of degarelix 80 mg per month at a concentration of 20 mg/mL (4 mL) at Days 28 to 168 were administered.
  During Phase B of the trial, If a patient had Prostate Specific Antigen (PSA) ≥2 ng/mL at any visit, additional doses of degarelix 240 mg followed by 80 mg maintenance dose(s) were administered.
  Interventions: Drug: Degarelix
- DC (Degarelix Continuous) (Experimental): Patients in this arm received degarelix with a starting dose of 240 mg at a concentration of 40 mg/mL administered on Day 0 (Visit 1) s.c. into the anterior abdominal wall via two equivalent injections of 120 mg (3 mL) each.
  Thirteen maintenance doses of degarelix 80 mg per month at a concentration of 20 mg/mL (4 mL) at Days 28 to 364, administered s.c. into the anterior abdominal wall
  Interventions: Drug: Degarelix
- LC (Leuprolide Continuous) (Active Comparator): Patients in this arm received leuprolide 7.5 mg one-month depot injection on Day 0, administered intramuscular (i.m.) into a large muscle, as per manufacturer's labeling directions.
  One injection of 22.5 mg leuprolide 3-month depot was administered i.m. as per manufacturer's labeling directions at Day 28 and every 3 months afterwards for 4 additional doses (i.e at Days 112, 196, 280, and 364, respectively).
  On Investigator's discretion, patients in the arm could take bicalutamide (Casodex®) for a maximum of 28 days to alleviate increased signs and symptoms due to initial upsurge in testosterone levels.
  Interventions: Drug: Leuprolide

INTERVENTIONS:
Drug: Degarelix — Degarelix treatment provided for first seven months (one starting dose and six maintenance doses) followed by no treatment for next seven months period.
  Arms: DI (Degarelix Intermittent)
Drug: Degarelix — Degarelix treatment provided for complete study period (one starting dose and 13 maintenance doses).
  Arms: DC (Degarelix Continuous)
Drug: Leuprolide — Leuprolide treatment for complete study period (one starting dose and 5 maintenance doses of 3-month depot each)
  Arms: LC (Leuprolide Continuous)

SUMMARY:
The purpose of this study was to see if giving Degarelix every month for 7 months then stop treatment for 7 months (intermittent therapy) would show a reduction of negative effects of androgen deprivation therapy by increasing the quality of life while keeping prostate specific antigen (PSA) levels suppressed.

DETAILED DESCRIPTION:
This was an open-label, randomized, parallel-arm, multicenter study to determine if degarelix intermittent therapy was non-inferior to continuous androgen deprivation therapy (combination of treatment groups receiving continuous degarelix and leuprolide therapy, respectively) in maintaining PSA levels at ≤ 4.0 ng/mL at 14 months.

The study consisted of two phases, Phase A and B. During Phase A, patients in the degarelix intermittent and degarelix continuous arms received 7 months of therapy with degarelix one-month depot formulation and patients in the leuprolide continuous arm received leuprolide one-month depot injection (7.5 mg) followed by two 3-month depot (22.5 mg) injections. After 7 months of treatment, patients with a PSA ≤2 ng/mL continued into Phase B.

During Phase B, patients in the degarelix intermittent arm had a 7-month off-treatment period. Patients randomized to the degarelix continuous arm and the leuprolide continuous arm continued to receive degarelix or leuprolide depot as in Phase A for the remainder of the 14 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Raising PSA after prior treatment failure of localized prostate cancer.
* Has a histological confirmed non-metastatic cancer of the prostate (Gleason graded) based on the most current biopsy.
* Has a screening testosterone within normal range (≥1.5 ng/mL).
* Has Eastern Cooperative Oncology Group score of ≤2.
* Bone scan or CT scan report documenting no evidence of metastasis to the bone or internal organs.
* Life expectancy of at least 15 months.

Exclusion Criteria:

* Taken hormone therapy in the last 6 months prior to entering this study.
* Being treated with 5-alpha reductase inhibitor at time of enrolment and remained on a stable dose throughout the trial.
* Has a history of severe uncontrolled asthma, anaphylactic reactions, or severe urticaria and/or angioedema.
* Has hypersensitivity towards any component of the study drug.
* Has a previous history or presence of another malignancy other than prostate cancer or treated squamous/basal cell carcinoma of the skin within the last five years.
* Has abnormal laboratory results which in the judgement of the Investigator would affect the patient's health or the outcome of the trial.
* Has a clinically significant medical condition (other than prostate cancer) including but not limited to; renal, haematological, gastrointestinal, endocrine, cardiac, neurological or psychiatric disease and alcohol or drug abuse or any other condition which may affect the patient's health or the outcome of the trial as judged by the Investigator.
* Has an intellectual incapacity or language barriers precluding adequate understanding or co-operation.
* Has received an investigational drug within the last 28 days before the Screening visit or longer if considered to possibly influence the outcome of the current trial.
* Has received ketoconazole or diflucan in the last 28 days preceding the Screening Visit.
* Has previously participated in any Degarelix trial.
* Is part of an ongoing trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2009-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (59):
- United States (59):
  - Alabama Clinical Research, Inc, Alexander City, Alabama
  - Urology Center of Alabama, PC, Homewood, Alabama
  - Advanced Urology Medical Center, Anaheim, California
  - Peninsula Urology Medical Center, Atherton, California
  - Urology Associates of Central California, Fresno, California
  - South Orange County Medical Research Center, Laguna Hills, California
  - Atlantic Urology Medical Group, Long Beach, California
  - San Bernardino Urological Associates, San Bernardino, California
  - San Diego Uro-Research, San Diego, California
  - Santa Barbara Clinical Research, Santa Barbara, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - The Urology Center of Colorado, Denver, Colorado
  - Urology Associates Research, Englewood, Colorado
  - Connecticut Clinical Research Center, Middlebury, Connecticut
  - Grove Hill Medical Center, New Britain, Connecticut
  - Walter Reed Army Hospital Medical Center, Washington D.C., District of Columbia
  - South Florida Medical Research, Aventura, Florida
  - Urology Health Solutions, Inc, Celebration, Florida
  - Florida Urology Physicians, Fort Myers, Florida
  - University of Florida, Gainesville, Florida
  - Winter Park Urology Associates, Orlando, Florida
  - Southeastern Urology Center, PA, Tallahassee, Florida
  - Tampa Bay Urology, Tampa, Florida
  - Advanced Research Institute, Inc, Trinity, Florida
  - Urology Enterprises, Marietta, Georgia
  - Midwest Urology/RMD Clinical Research Institute, Melrose Park, Illinois
  - Deaconess Clinic Inc, Evansville, Indiana
  - Northeast Indiana Research, Fort Wayne, Indiana
  - Metropolitan Urology, PSC, Jeffersonville, Indiana
  - Regional Urology, Lic, Shreveport, Louisiana
  - Chesapeake Urology Associates, Baltimore, Maryland
  - Chesapeake Urology Research Associates, Baltimore, Maryland
  - Chesapeake Urology Research Associates, Glen Burnie, Maryland
  - Myron Murdock M.D. LLC, Greenbelt, Maryland
  - Chesapeake Urology Associates, PA, Towson, Maryland
  - Urology Associates of Englewood, Englewood, New Jersey
  - Hamilton Urology PA, Hamilton, New Jersey
  - Lawrenceville Urology, Lawrenceville, New Jersey
  - Nationsmed Clinical Research, Perth Amboy, New Jersey
  - Center for Urologic Care, Voorhees Township, New Jersey
  - Delaware Valley Urology LLC, Woodlane, New Jersey
  - The Urological Institute of NE NY, CCP, Albany, New York
  - Medical & Clinical Research Associates, Bay Shore, New York
  - Brooklyn Heights Urology Associates, P.C., Brooklyn, New York
  - University Urology Associates, New York, New York
  - Hudson Valley Urology P.C., Poughkeepsie, New York
  - Northeast Urology Research, Concord, North Carolina
  - Alliance Urology Specialists, Greensboro, North Carolina
  - Urological Association of Lancaster, Lancaster, Pennsylvania
  - State College Urologic Association, State College, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Lexington Urological Associates, PA, West Columbia, South Carolina
  - Urology Associates, Nashville, Tennessee
  - Lackland Air Force base, San Antonio, Texas
  - Urology of Virginia, Norfolk, Virginia
  - Virginal Urology, Richmond, Virginia
  - Virginia Urology Center, Richmond, Virginia
  - Seattle Urology Research Center, Seattle, Washington
  - Roger D. Fincher, PS, Spokane, Washington

REFERENCES:
- [Derived] Zengerling F, Jakob JJ, Schmidt S, Meerpohl JJ, Blumle A, Schmucker C, Mayer B, Kunath F. Degarelix for treating advanced hormone-sensitive prostate cancer. Cochrane Database Syst Rev. 2021 Aug 5;8(8):CD012548. doi: 10.1002/14651858.CD012548.pub2. PMID 34350976

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the total 409 patients enrolled, six patients were not dosed either due to randomisation error, failing eligibility criteria or consent withdrawal after being randomised.
Groups:
- DI (Degarelix Intermittent): Patients in this arm received degarelix with a starting dose of 240 mg at a concentration of 40 mg/mL on Day 0 (Visit 1) administered subcutaneously (s.c.) into the anterior abdominal wall via two equivalent injections of 120 mg (3 mL) each.
  Six maintenance doses of degarelix 80 mg per month at a concentration of 20 mg/mL (4 mL) at Days 28 to 168 (Visit 2 through 7), administered s.c. into the anterior abdominal wall
  During Phase B of the trial, If a patient had Prostate Specific Antigen (PSA) ≥2 ng/mL at any visit, additional doses of degarelix 240 mg followed by 80 mg maintenance dose(s) were administered.
  Degarelix: Degarelix treatment provided for first seven months (one starting dose and six maintenance doses) followed by no treatment for next seven months period.
- DC (Degarelix Continuous): Patients in this arm received degarelix with a starting dose of 240 mg at a concentration of 40 mg/mL administered on Day 0 (Visit 1) s.c. into the anterior abdominal wall via two equivalent injections of 120 mg (3 mL) each.
  Thirteen maintenance doses of degarelix 80 mg per month at a concentration of 20 mg/mL (4 mL) at Days 28 to 364, administered s.c. into the anterior abdominal wall
  Degarelix: Degarelix treatment provided for complete study period (one starting dose and 13 maintenance doses).
- LC (Leuprolide Continuous): Patients in this arm received leuprolide 7.5 mg one-month depot injection on Day 0 (Visit 1), administered intramuscular (i.m.) into a large muscle, as per manufacturer's labeling directions.
  One injection of 22.5 mg leuprolide 3-month depot was administered i.m. into a large muscle, according to the directions for use in the manufacturer's labeling at Day 28 and every 3 months afterwards for 4 additional doses (i.e at Days 112, 196, 280, and 364, respectively).
  On Investigator's discretion, patients in the arm could take bicalutamide (Casodex®) for a maximum of 28 days to alleviate increased signs and symptoms due to initial upsurge in testosterone levels.
  Leuprolide: Leuprolide treatment for complete study period (one starting dose and 5 maintenance doses of 3-month depot each).
Period: Overall Study
Arm/Group | DI (Degarelix Intermittent) | DC (Degarelix Continuous) | LC (Leuprolide Continuous)
Started | 175 (Full Analysis Set Patients) | 50 (Full Analysis Set Patients) | 178 (Full Analysis Set Patients)
Full Phase B Analysis Set | 137 (Patients completing 7 months treatment with PSA<2 ng/mL, and having one primary efficacy assessment.) | 41 (Patients completing 7 months treatment with PSA<2 ng/mL, and having one primary efficacy assessment.) | 150 (Patients completing 7 months treatment with PSA<2 ng/mL, and having one primary efficacy assessment.)
Completed | 131 | 36 | 134
Not Completed | 44 | 14 | 44
Not completed — Adverse Event | 14 | 5 | 18
Not completed — Protocol Violation | 5 | 0 | 8
Not completed — Physician Decision | 2 | 0 | 3
Not completed — Lost to Follow-up | 1 | 0 | 3
Not completed — Withdrawal by Subject | 5 | 3 | 2
Not completed — PSA failure (>2 ng/mL) at Visit 8 | 10 | 4 | 7
Not completed — PSA failure (>2 ng/mL) on other visit | 2 | 1 | 1
Not completed — Other (not meeting above criteria) | 5 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Analysis population consist of Full Analysis Set (FAS), which comprised of subjects who received at least one dose of IMP and had at least one efficacy assessment after dosing.
Groups:
- DI (Degarelix Intermittent): Patients in this arm received degarelix with a starting dose of 240 mg at a concentration of 40 mg/mL on Day 0 administered subcutaneously (s.c.) into the anterior abdominal wall via two equivalent injections of 120 mg (3 mL) each.
  Six maintenance doses of degarelix 80 mg per month at a concentration of 20 mg/mL (4 mL) at Days 28 to 168 were administered.
  During Phase B of the trial, If a patient had Prostate Specific Antigen (PSA) ≥2 ng/mL at any visit, additional doses of degarelix 240 mg followed by 80 mg maintenance dose(s) were administered.
  Degarelix: Degarelix treatment provided for first seven months (one starting dose and six maintenance doses) followed by no treatment for next seven months period.
- LC (Leuprolide Continuous): Patients in this arm received leuprolide 7.5 mg one-month depot injection on Day 0, administered intramuscular (i.m.) into a large muscle, as per manufacturer's labeling directions.
  One injection of 22.5 mg leuprolide 3-month depot was administered i.m. as per manufacturer's labeling directions at Day 28 and every 3 months afterwards for 4 additional doses (i.e at Days 112, 196, 280, and 364, respectively).
  On Investigator's discretion, patients in the arm could take bicalutamide (Casodex®) for a maximum of 28 days to alleviate increased signs and symptoms due to initial upsurge in testosterone levels.
  Leuprolide: Leuprolide treatment for complete study period (one starting dose and 5 maintenance doses of 3-month depot each)
- Total: Total of all reporting groups
Arm/Group | DI (Degarelix Intermittent) | DC (Degarelix Continuous) | LC (Leuprolide Continuous) | Total
Number analyzed (Participants) | 175 | 50 | 178 | 403
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.9 (8.89) | 71.7 (8.14) | 71.0 (8.44) | 71.5 (8.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 175 | 50 | 178 | 403
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 4 | 14 | 35
  Not Hispanic or Latino | 158 | 46 | 164 | 368
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 2 | 5
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 32 | 9 | 38 | 79
  White | 140 | 39 | 137 | 316
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Height [Mean (Standard Deviation); unit: Meter] | 1.77 (0.089) | 1.74 (0.089) | 1.76 (0.080) | 1.76 (0.085)
Weight [Mean (Standard Deviation); unit: Kg] | 90.3 (19.4) | 88.4 (15.8) | 91.9 (16.9) | 90.8 (17.9)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] | 28.9 (5.45) | 29.2 (4.89) | 29.6 (4.94) | 29.2 (5.16)
Prostate Specific Antigen (PSA) [Mean (Standard Deviation); unit: ng/mL] | 16.4 (66.3) | 15.6 (32.2) | 10.7 (24.4) | 13.8 (48)
Testosterone [Mean (Standard Deviation); unit: ng/mL] | 3.65 (1.43) | 3.90 (1.59) | 3.76 (1.58) | 3.73 (1.52)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Serum PSA Levels ≤4.0 ng/mL
Description: Percentage of patients with serum PSA levels ≤4.0 ng/mL at 14 month was presented.
Time Frame: At 14 month
Population: Analysis set consist of Full Phase B Analysis Set, which comprised of patients who completed 7 months of treatment and had a PSA ≤2.0 ng/mL at the end of Month 7 and had at least one primary endpoint efficacy assessment after Month 7.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Groups:
- Total Continuous: This is the combination of degarelix continuous and leuprolide continuous treatment arms.
Arm/Group | DI (Degarelix Intermittent) | Total Continuous
Number analyzed (Participants) | 137 | 191
Percentage of patients | 100 [97.3 to 100] | 98.4 [95.5 to 99.7]
Statistical Analysis 1: Comparison: DI (Degarelix Intermittent) vs Total Continuous; Test type: Non-Inferiority or Equivalence — Non-inferiority was defined as a lower bound (LCL) of the 95% confidence interval for the difference between the intermittent and pooled continuous treatments, CADT, (intermittent - continuous) of greater than -12.5%; Percentage difference = 1.57, 95% CI 2-sided [-0.19 to 3.33]

2. Secondary Outcome: Absolute Change From Baseline in Serum PSA Levels
Description: Absolute change from Baseline in serum PSA levels during the study period was measured.
Time Frame: Phase A Visit 1-8 and Phase B Visit 9-15.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- DI (Degarelix Intermittent): Patients in this arm received degarelix with a starting dose of 240 mg at a concentration of 40 mg/mL on Day 0 (Visit 1) administered subcutaneously (s.c.) into the anterior abdominal wall via two equivalent injections of 120 mg (3 mL) each.
  Six maintenance doses of degarelix 80 mg per month at a concentration of 20 mg/mL (4 mL) at Days 28 to 168 (Visit 2 through 7), administered s.c. into the anterior abdominal wall.
  During Phase B of the trial, If a patient had Prostate Specific Antigen (PSA) ≥2 ng/mL at any visit, additional doses of degarelix 240 mg followed by 80 mg maintenance dose(s) were administered.
  Degarelix: Degarelix treatment provided for first seven months (one starting dose and six maintenance doses) followed by no treatment for next seven months period.
Arm/Group | DI (Degarelix Intermittent) | DC (Degarelix Continuous) | LC (Leuprolide Continuous)
Number analyzed (Participants) | 137 | 41 | 150
ng/mL
  Phase A, Visit 1 (Day 0) | NA (NA) — This visit was the first dosing visit. Serum samples were collected pre-dosing on this visit. Thus, the estimated value obtained on this visit were considered as Baseline value. Hence no change is reported. | -0.91 (NA) — One patient erroneously received medication prior to this visit. Thus, the value obtained on this visit was considered as first post-baseline value for this patient and is reported. There was no SD. | NA (NA) — This visit was the first dosing visit. Serum samples were collected pre-dosing on this visit. Thus, the estimated value obtained on this visit were considered as Baseline value. Hence no change is reported.
  Phase A, Visit 2 (Month 1) | -6.39 (10.2) | -14.3 (34.8) | -6.38 (13.2)
  Phase A, Visit 3 (Month 2) | -6.94 (10.8) | -14.8 (34.9) | -8.12 (15.4)
  Phase A, Visit 4 (Month 3) | -7.07 (10.9) | -15 (35) | -8.44 (15.7)
  Phase A, Visit 5 (Month 4) | -7.16 (11) | -15.1 (35.2) | -8.51 (15.8)
  Phase A, Visit 6 (Month 5) | -7.19 (11) | -15.1 (35.2) | -8.59 (15.9)
  Phase A, Visit 7 (Month 6) | -7.21 (10.9) | -15.1 (35.2) | -8.64 (15.9)
  Phase A, Visit 8 (Month 7) | -7.24 (11) | -15.1 (35.2) | -8.64 (15.9)
  Phase B, Visit 9 (Month 8) | -7.25 (11) | -15 (34.7) | -8.64 (15.9)
  Phase B, Visit 10 (Month 9) | -7.18 (11) | -15 (34.7) | -8.64 (15.9)
  Phase B, Visit 11 (Month 10) | -7.07 (10.9) | -14.9 (34.3) | -8.63 (15.9)
  Phase B, Visit 12 (Month 11) | -6.96 (10.9) | -14.9 (33.9) | -8.64 (15.9)
  Phase B, Visit 13 (Month 12) | -6.81 (11) | -14.8 (33.9) | -8.64 (15.9)
  Phase B, Visit 14 (Month 13) | -6.79 (11) | -14.8 (33.9) | -8.59 (16)
  Phase B, Visit 15 (Month 14) | -6.74 (11) | -14.8 (33.9) | -8.6 (15.9)

3. Secondary Outcome: Percent Change From Baseline in Serum PSA Levels
Description: Percent change from Baseline in serum PSA levels during the study period was measured.
Time Frame: Phase A Visit 1-8 and Phase B Visit 9-15.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | DI (Degarelix Intermittent) | DC (Degarelix Continuous) | LC (Leuprolide Continuous)
Number analyzed (Participants) | 137 | 41 | 150
Percent change
  Phase A, Visit 1 (Day 0) | NA (NA) — This visit was the first dosing visit. Serum samples were collected pre-dosing on this visit. Thus, the estimated value obtained on this visit were considered as Baseline value. Hence no change is reported. | -39.6 (NA) — One patient erroneously received medication prior to this visit. Thus, the value obtained on this visit was considered as first post-baseline value for this patient and is reported. There was no SD. | NA (NA) — This visit was the first dosing visit. Serum samples were collected pre-dosing on this visit. Thus, the estimated value obtained on this visit were considered as Baseline value. Hence no change is reported.
  Phase A, Visit 2 (Month 1) | -80.8 (24.4) | -84.5 (11.8) | -62.8 (31.2)
  Phase A, Visit 3 (Month 2) | -90.4 (12.2) | -92.4 (8.23) | -87.3 (12.3)
  Phase A, Visit 4 (Month 3) | -92.8 (9.9) | -94.5 (7.37) | -92.3 (7.67)
  Phase A, Visit 5 (Month 4) | -94.1 (8.45) | -95.5 (7.05) | -93.4 (9.39)
  Phase A, Visit 6 (Month 5) | -94.2 (9.31) | -95.7 (7.8) | -94.5 (7.52)
  Phase A, Visit 7 (Month 6) | -94.8 (8.34) | -95.8 (8.64) | -95.3 (7.23)
  Phase A, Visit 8 (Month 7) | -95.4 (7.13) | -95.4 (10.8) | -95.5 (7.62)
  Phase B, Visit 9 (Month 8) | -95.7 (6.97) | -95.5 (10.3) | -95.2 (12.3)
  Phase B, Visit 10 (Month 9) | -93.6 (11.5) | -95.6 (10.6) | -94.3 (23.2)
  Phase B, Visit 11 (Month 10) | -91.9 (13.4) | -95.7 (9.46) | -93.1 (24.9)
  Phase B, Visit 12 (Month 11) | -88 (22.7) | -95.1 (11.9) | -94.4 (23.5)
  Phase B, Visit 13 (Month 12) | -84.2 (24.9) | -95.1 (10.6) | -94.5 (23.5)
  Phase B, Visit 14 (Month 13) | -82.8 (24.9) | -95.1 (10.4) | -93.1 (25.9)
  Phase B, Visit 15 (Month 14) | -80.8 (26.4) | -94.4 (12.9) | -93.7 (25.8)

4. Secondary Outcome: Change From Baseline in Quality of Life as Assessed by the Functional Assessment of Cancer Therapy-Prostate (FACT-P) : Physical Well-being
Description: The FACT-P is a multidimensional, self-report quality of life (QoL) instrument specifically designed for use with prostate cancer patients. It consists of 27 core items which assess patient function in four domains: Physical, Social/Family, Emotional, and Functional well-being, which is further supplemented by 12 site specific items to assess for prostate related symptoms. Each question is rated on a scale from 0 to 4, and then combined to produce sub-scale scores for each domain, as well as a global QoL score.
  Physical well-being consist of 7 items and scored on a scale of 0-4 (0=Not at all; 1=A little bit; 2=Somewhat; 3=Quite a bit; 4=Very much). Total score for the physical well-being sub scale ranges from 0 to 28. Higher scores represent better QoL.
Time Frame: During 14 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Groups:
- LC (Leuprolide Continuous): Patients in this arm received leuprolide 7.5 mg one-month depot injection on Day 0 (Visit 1), administered intramuscular (i.m.) into a large muscle, as per manufacturer's labeling directions.
  One injection of 22.5 mg leuprolide 3-month depot was administered i.m. into a large muscle, according to the directions for use in the manufacturer's labeling at Day 28 and every 3 months afterwards for 4 additional doses (i.e at Days 112, 196, 280, and 364, respectively).
  On Investigator's discretion, patients in the arm could take bicalutamide (Casodex®) for a maximum of 28 days to alleviate increased signs and symptoms due to initial upsurge in testosterone levels.
  Leuprolide: Leuprolide treatment for complete study period (one starting dose and 5 maintenance doses of 3- month depot each).
Arm/Group | DI (Degarelix Intermittent) | DC (Degarelix Continuous) | LC (Leuprolide Continuous) | Total Continuous
Number analyzed (Participants) | 137 | 41 | 150 | 191
Scores on a scale
  Phase A, Month 3 | -1.47 [-1.99 to -0.94] | -1.63 [-2.59 to -0.67] | -1.41 [-1.92 to -0.90] | -1.46 [-1.90 to -1.01]
  Phase A, Month 7 | -1.41 [-1.93 to -0.88] | -1.48 [-2.43 to -0.52] | -1.67 [-2.17 to -1.17] | -1.63 [-2.07 to -1.18]
  Phase B, Month 8 | -0.96 [-1.46 to -0.46] | -1.92 [-2.83 to -1.01] | -1.74 [-2.22 to -1.27] | -1.78 [-2.20 to -1.36]
  Phase B, Month 9 | -1.24 [-1.80 to -0.68] | -1.85 [-2.87 to -0.82] | -1.77 [-2.31 to -1.24] | -1.79 [-2.26 to -1.32]
  Phase B, Month 10 | -1.05 [-1.63 to -0.48] | -2.08 [-3.13 to -1.03] | -1.68 [-2.23 to -1.13] | -1.76 [-2.25 to -1.28]
  Phase B, Month 11 | -1.00 [-1.56 to -0.44] | -1.77 [-2.79 to -0.75] | -1.53 [-2.07 to -1.00] | -1.58 [-2.05 to -1.11]
  Phase B, Month 12 | -0.91 [-1.44 to -0.38] | -1.62 [-2.59 to -0.66] | -1.32 [-1.83 to -0.82] | -1.39 [-1.83 to -0.94]
  Phase B, Month 13 | -1.00 [-1.57 to -0.43] | -2.10 [-3.14 to -1.06] | -1.40 [-1.95 to -0.86] | -1.55 [-2.04 to -1.07]
  Phase B, Month 14 | -1.04 [-1.62 to -0.47] | -1.90 [-2.95 to -0.85] | -1.45 [-2.00 to -0.91] | -1.55 [-2.03 to -1.06]

5. Secondary Outcome: Change From Baseline in Quality of Life as Assessed by the FACT-P : Emotional Well-being
Description: The FACT-P is a multidimensional, self-report quality of life (QoL) instrument specifically designed for use with prostate cancer patients. It consists of 27 core items which assess patient function in four domains: Physical, Social/Family, Emotional, and Functional well-being, which is further supplemented by 12 site specific items to assess for prostate related symptoms. Each question is rated on a scale from 0 to 4, and then combined to produce sub-scale scores for each domain, as well as a global QoL score.
  Emotional well-being consist of 6 items and scored on a scale of 0-4 (0=Not at all; 1=A little bit; 2=Somewhat; 3=Quite a bit; 4=Very much). Total score for the emotional well-being sub scale ranges from 0 to 24. Higher scores represent better QoL.Higher scores represent better QoL.
Time Frame: During 14 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Groups:
- DC (Degarelix Continuous): administered on Day 0 (Visit 1) s.c. into the anterior abdominal wall via two equivalent injections of 120 mg (3 mL) each.
  Thirteen maintenance doses of degarelix 80 mg per month at a concentration of 20 mg/mL (4 mL) at Days 28 to 364, administered s.c. into the anterior abdominal wall.
  Degarelix: Degarelix treatment provided for complete study period (one starting dose and 13 maintenance doses).
Arm/Group | DI (Degarelix Intermittent) | DC (Degarelix Continuous) | LC (Leuprolide Continuous) | Total Continuous
Number analyzed (Participants) | 137 | 41 | 150 | 191
Scores on a scale
  Phase A, Month 3 | 0.69 [0.18 to 1.20] | 1.31 [0.37 to 2.24] | 0.76 [0.27 to 1.24] | 0.88 [0.45 to 1.30]
  Phase A, Month 7 | 0.67 [0.16 to 1.18] | 0.57 [-0.37 to 1.51] | 0.90 [0.42 to 1.39] | 0.83 [0.40 to 1.26]
  Phase B, Month 8 | 0.65 [0.16 to 1.14] | 0.95 [0.05 to 1.86] | 1.11 [0.65 to 1.58] | 1.08 [0.67 to 1.49]
  Phase B, Month 9 | 0.75 [0.27 to 1.24] | 1.11 [0.22 to 2.01] | 1.16 [0.70 to 1.62] | 1.15 [0.74 to 1.56]
  Phase B, Month 10 | 1.09 [0.57 to 1.60] | 0.00 [-0.94 to 0.95] | 0.98 [0.49 to 1.46] | 0.77 [0.34 to 1.20]
  Phase B, Month 11 | 0.82 [0.34 to 1.30] | 0.94 [0.06 to 1.83] | 1.05 [0.59 to 1.50] | 1.03 [0.62 to 1.43]
  Phase B, Month 12 | 0.99 [0.47 to 1.50] | 1.07 [0.12 to 2.02] | 1.23 [0.74 to 1.72] | 1.20 [0.76 to 1.63]
  Phase B, Month 13 | 0.74 [0.22 to 1.26] | 0.52 [-0.43 to 1.48] | 1.14 [0.64 to 1.63] | 1.01 [0.57 to 1.45]
  Phase B, Month 14 | 0.40 [-0.13 to 0.93] | 0.86 [-0.11 to 1.83] | 1.12 [0.62 to 1.62] | 1.06 [0.62 to 1.51]

6. Secondary Outcome: Change From Baseline in Quality of Life as Assessed by the FACT-P : Social Well-being
Description: The FACT-P is a multidimensional, self-report quality of life (QoL) instrument specifically designed for use with prostate cancer patients. It consists of 27 core items which assess patient function in four domains: Physical, Social/Family, Emotional, and Functional well-being, which is further supplemented by 12 site specific items to assess for prostate related symptoms. Each question is rated on a scale from 0 to 4, and then combined to produce sub-scale scores for each domain, as well as a global QoL score.
  Social well-being consist of 7 items and scored on a scale of 0-4 (0=Not at all; 1=A little bit; 2=Somewhat; 3=Quite a bit; 4=Very much). Total score for the social well-being sub scale ranges from 0 to 28. Higher scores represent better QoL.
Time Frame: During 14 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Groups:
- DC (Degarelix Continuous): Patients in this arm received degarelix with a starting dose of 240 mg at a concentration of 40 mg/mL administered on Day 0 (Visit 1) s.c. into the anterior abdominal wall via two equivalent injections of 120 mg (3 mL) each.
  Thirteen maintenance doses of degarelix 80 mg per month at a concentration of 20 mg/mL (4 mL) at Days 28 to 364, administered s.c. into the anterior abdominal wall.
  Degarelix: Degarelix treatment provided for complete study period (one starting dose and 13 maintenance doses).
Arm/Group | DI (Degarelix Intermittent) | DC (Degarelix Continuous) | LC (Leuprolide Continuous) | Total Continuous
Number analyzed (Participants) | 137 | 41 | 150 | 191
Scores on a scale
  Phase A, Month 3 | -0.18 [-0.96 to 0.60] | -0.06 [-1.48 to 1.35] | -0.36 [-1.11 to 0.38] | -0.30 [-0.95 to 0.36]
  Phase A, Month 7 | 0.00 [-0.79 to 0.79] | -0.30 [-1.75 to 1.14] | -0.46 [-1.21 to 0.29] | -0.43 [-1.09 to 0.24]
  Phase B, Month 8 | -0.33 [-1.06 to 0.39] | -0.52 [-1.84 to 0.80] | -0.41 [-1.10 to 0.28] | -0.43 [-1.04 to 0.18]
  Phase B, Month 9 | -0.02 [-0.80 to 0.77] | -0.95 [-2.37 to 0.47] | -1.10 [-1.84 to -0.36] | -1.07 [-1.72 to -0.41]
  Phase B, Month 10 | 0.36 [-0.42 to 1.14] | -1.00 [-2.42 to 0.42] | -1.15 [-1.89 to -0.41] | -1.12 [-1.77 to -0.46]
  Phase B, Month 11 | 0.20 [-0.63 to 1.02] | -1.09 [-2.59 to 0.42] | -0.83 [-1.61 to -0.05] | -0.88 [-1.58 to -0.19]
  Phase B, Month 12 | -0.16 [-0.94 to 0.63] | -1.34 [-2.78 to 0.09] | -0.85 [-1.59 to -0.10] | -0.95 [-1.61 to -0.29]
  Phase B, Month 13 | -0.02 [-0.79 to 0.74] | -1.35 [-2.74 to 0.03] | -0.72 [-1.44 to 0.00] | -0.85 [-1.49 to -0.21]
  Phase B, Month 14 | 0.28 [-0.44 to 1.01] | -0.68 [-2.00 to 0.64] | -0.55 [-1.24 to 0.14] | -0.58 [-1.19 to 0.03]

7. Secondary Outcome: Change From Baseline in Quality of Life as Assessed by the FACT-P : Functional Well-being
Description: The FACT-P is a multidimensional, self-report quality of life (QoL) instrument specifically designed for use with prostate cancer patients. It consists of 27 core items which assess patient function in four domains: Physical, Social/Family, Emotional, and Functional well-being, which is further supplemented by 12 site specific items to assess for prostate related symptoms. Each question is rated on a scale from 0 to 4, and then combined to produce sub-scale scores for each domain, as well as a global QoL score.
  Functional well-being consist of 7 items and scored on a scale of 0-4 (0=Not at all; 1=A little bit; 2=Somewhat; 3=Quite a bit; 4=Very much). Total score for the functional well-being sub scale ranges from 0 to 28. Higher scores represent better QoL.
Time Frame: During 14 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | DI (Degarelix Intermittent) | DC (Degarelix Continuous) | LC (Leuprolide Continuous) | Total Continuous
Number analyzed (Participants) | 137 | 41 | 150 | 191
Scores on a scale
  Phase A, Month 3 | -0.96 [-1.70 to -0.23] | -0.88 [-2.23 to 0.47] | -0.29 [-0.99 to 0.41] | -0.42 [-1.04 to 0.21]
  Phase A, Month 7 | -1.41 [-2.25 to -0.58] | -0.78 [-2.31 to 0.76] | -1.24 [-2.03 to -0.45] | -1.15 [-1.85 to -0.44]
  Phase B, Month 8 | -1.18 [-1.90 to -0.45] | -1.08 [-2.41 to 0.26] | -0.73 [-1.42 to -0.04] | -0.80 [-1.41 to -0.19]
  Phase B, Month 9 | -1.14 [-1.94 to -0.34] | -1.07 [-2.53 to 0.40] | -1.23 [-1.99 to -0.47] | -1.20 [-1.87 to -0.52]
  Phase B, Month 10 | -1.35 [-2.15 to -0.54] | -0.89 [-2.36 to 0.58] | -1.42 [-2.18 to -0.66] | -1.31 [-1.98 to -0.63]
  Phase B, Month 11 | -1.25 [-2.08 to -0.43] | -0.80 [-2.32 to 0.72] | -1.24 [-2.02 to -0.46] | -1.15 [-1.84 to -0.45]
  Phase B, Month 12 | -0.92 [-1.70 to -0.15] | -1.49 [-2.91 to -0.07] | -0.73 [-1.46 to 0.00] | -0.89 [-1.54 to -0.24]
  Phase B, Month 13 | -1.49 [-2.32 to -0.66] | -2.22 [-3.75 to -0.69] | -0.96 [-1.75 to -0.17] | -1.22 [-1.93 to -0.52]
  Phase B, Month 14 | -1.02 [-1.78 to -0.26] | -1.95 [-3.35 to -0.55] | -0.84 [-1.56 to -0.12] | -1.07 [-1.71 to -0.43]

8. Secondary Outcome: Change From Baseline in Quality of Life as Assessed by the FACT-P : Additional Concerns
Description: The FACT-P is a multidimensional, self-report quality of life (QoL) instrument specifically designed for use with prostate cancer patients. It consists of 27 core items which assess patient function in four domains: Physical, Social/Family, Emotional, and Functional well-being, which is further supplemented by 12 site specific items to assess for prostate related symptoms. Each question is rated on a scale from 0 to 4, and then combined to produce sub-scale scores for each domain, as well as a global QoL score.
  Additional concerns consist of 12 items and scored on a scale of 0-4 (0=Not at all; 1=A little bit; 2=Somewhat; 3=Quite a bit; 4=Very much). Total score for the additional concerns ranges from 0 to 48. Higher scores represent better QoL.
Time Frame: During 14 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | DI (Degarelix Intermittent) | DC (Degarelix Continuous) | LC (Leuprolide Continuous) | Total Continuous
Number analyzed (Participants) | 137 | 41 | 150 | 191
Scores on a scale
  Phase A, Month 3 | -1.14 [-1.96 to -0.32] | -0.92 [-2.42 to 0.57] | -0.51 [-1.30 to 0.27] | -0.60 [-1.29 to 0.09]
  Phase A, Month 7 | -0.89 [-1.71 to -0.07] | -1.34 [-2.83 to 0.16] | -1.03 [-1.81 to -0.25] | -1.10 [-1.79 to -0.40]
  Phase B, Month 8 | -1.29 [-2.10 to -0.48] | -1.03 [-2.50 to 0.45] | -0.63 [-1.40 to 0.14] | -0.72 [-1.40 to -0.03]
  Phase B, Month 9 | -0.97 [-1.83 to -0.11] | -1.64 [-3.20 to -0.07] | -0.90 [-1.72 to -0.08] | -1.06 [-1.79 to -0.34]
  Phase B, Month 10 | -0.86 [-1.73 to 0.01] | -0.80 [-2.39 to 0.78] | -0.70 [-1.52 to 0.13] | -0.72 [-1.45 to 0.01]
  Phase B, Month 11 | -0.80 [-1.62 to 0.01] | -0.56 [-2.05 to 0.92] | -0.58 [-1.35 to 0.20] | -0.57 [-1.26 to 0.11]
  Phase B, Month 12 | -0.75 [-1.60 to 0.10] | -1.20 [-2.75 to 0.35] | -0.75 [-1.56 to 0.06] | -0.84 [-1.56 to -0.13]
  Phase B, Month 13 | -0.91 [-1.75 to -0.08] | -0.96 [-2.47 to 0.56] | -0.86 [-1.65 to -0.06] | -0.88 [-1.58 to -0.18]
  Phase B, Month 14 | -0.81 [-1.69 to 0.06] | -0.67 [-2.26 to 0.92] | -0.27 [-1.10 to 0.57] | -0.35 [-1.09 to 0.38]

9. Secondary Outcome: Change From Baseline in Quality of Life as Assessed by the FACT-P: Total FACT-P Score
Description: The FACT-P is a multidimensional, self-report quality of life (QoL) instrument specifically designed for use with prostate cancer patients. It consists of 27 core items which assess patient function in four domains: Physical, Social/Family, Emotional, and Functional well-being, which is further supplemented by 12 site specific items to assess for prostate related symptoms. Each question is rated on a scale from 0 to 4, and then combined to produce sub-scale scores for each domain, as well as a global QoL score. Total FACT-P scores ranges from 0 to 156. Higher scores represent better QoL.
Time Frame: During 14 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | DI (Degarelix Intermittent) | DC (Degarelix Continuous) | LC (Leuprolide Continuous) | Total Continuous
Number analyzed (Participants) | 137 | 41 | 150 | 191
Scores on a scale
  Phase A, Month 3 | -1.86 [-3.62 to -0.10] | -1.89 [-5.13 to 1.34] | -1.23 [-2.92 to 0.45] | -1.37 [-2.87 to 0.12]
  Phase A, Month 7 | -2.03 [-3.87 to -0.19] | -2.64 [-6.03 to 0.76] | -2.38 [-4.12 to -0.63] | -2.43 [-3.98 to -0.88]
  Phase B, Month 8 | -1.75 [-3.45 to -0.04] | -3.12 [-6.26 to 0.03] | -1.69 [-3.31 to -0.07] | -1.99 [-3.42 to -0.55]
  Phase B, Month 9 | -1.61 [-3.46 to 0.23] | -3.49 [-6.89 to -0.10] | -2.84 [-4.59 to -1.09] | -2.98 [-4.53 to -1.42]
  Phase B, Month 10 | -0.89 [-2.84 to 1.05] | -4.56 [-8.15 to -0.98] | -3.16 [-5.01 to -1.31] | -3.45 [-5.09 to -1.81]
  Phase B, Month 11 | -1.18 [-3.10 to 0.73] | -3.27 [-6.79 to 0.26] | -2.48 [-4.30 to -0.67] | -2.65 [-4.26 to -1.04]
  Phase B, Month 12 | -0.95 [-2.88 to 0.98] | -3.97 [-7.52 to -0.42] | -1.60 [-3.43 to 0.23] | -2.09 [-3.72 to -0.47]
  Phase B, Month 13 | -1.74 [-3.72 to 0.24] | -5.62 [-9.26 to -1.97] | -1.85 [-3.73 to 0.02] | -2.64 [-4.32 to -0.97]
  Phase B, Month 14 | -1.36 [-3.24 to 0.52] | -4.28 [-7.75 to -0.81] | -1.65 [-3.44 to 0.13] | -2.20 [-3.79 to -0.61]

10. Secondary Outcome: Change From Baseline in Sexual Function as Assessed by the Sexual Function Index (SFI): Sexual Drive
Description: The SFI is a multidimensional, self-report instrument specifically designed to evaluate sexual function and satisfaction of men on treatment or with conditions that may affect sexual function. It consists of 11 questions which assess patient function in four domains: Sexual drive, Erection, Ejaculation, and Problem assessment, and a question in regards to overall assessment of sexual function.
  Sexual drive domain consist of 2 questions and are scored on a scale of 0-4 (0=minimum, 4=maximum). Total score for the sexual drive domain ranges from 0 to 8. A higher scores represent better sexual function.
Time Frame: During 14 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | DI (Degarelix Intermittent) | DC (Degarelix Continuous) | LC (Leuprolide Continuous) | Total Continuous
Number analyzed (Participants) | 137 | 41 | 150 | 191
Scores on a scale
  Phase A, Month 3 | -1.57 [-1.83 to -1.32] | -1.57 [-2.04 to -1.10] | -1.27 [-1.51 to -1.03] | -1.33 [-1.55 to -1.12]
  Phase A, Month 7 | -1.71 [-1.96 to -1.47] | -1.39 [-1.84 to -0.94] | -1.67 [-1.90 to -1.44] | -1.61 [-1.82 to -1.41]
  Phase B, Month 9 | -1.72 [-1.98 to -1.46] | -1.51 [-1.99 to -1.02] | -1.62 [-1.87 to -1.37] | -1.60 [-1.82 to -1.38]
  Phase B, Month 11 | -1.59 [-1.85 to -1.34] | -1.52 [-1.99 to -1.05] | -1.65 [-1.89 to -1.42] | -1.63 [-1.84 to -1.41]
  Phase B, Month 13 | -1.44 [-1.69 to -1.19] | -1.55 [-2.02 to -1.08] | -1.72 [-1.96 to -1.48] | -1.69 [-1.90 to -1.47]
  Phase B, Month 14 | -1.30 [-1.55 to -1.04] | -1.65 [-2.12 to -1.17] | -1.72 [-1.96 to -1.48] | -1.71 [-1.92 to -1.49]

11. Secondary Outcome: Change From Baseline in Sexual Function as Assessed by the SFI: Erection
Description: The SFI is a multidimensional, self-report instrument specifically designed to evaluate sexual function and satisfaction of men on treatment or with conditions that may affect sexual function. It consists of 11 questions which assess patient function in four domains: Sexual drive, Erection, Ejaculation, and Problem assessment, and a question in regards to overall assessment of sexual function.
  Erection domain consist of 3 questions and are scored on a scale of 0-4 (0=minimum, 4=maximum). Total score for the erection domain ranges from 0 to 12. A higher scores represent better sexual function.
Time Frame: During 14 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | DI (Degarelix Intermittent) | DC (Degarelix Continuous) | LC (Leuprolide Continuous) | Total Continuous
Number analyzed (Participants) | 137 | 41 | 150 | 191
Scores on a scale
  Phase A, Month 3 | -1.32 [-1.62 to -1.01] | -0.91 [-1.48 to -0.35] | -1.21 [-1.50 to -0.91] | -1.14 [-1.40 to -0.89]
  Phase A, Month 7 | -1.43 [-1.75 to -1.11] | -1.06 [-1.65 to -0.47] | -1.34 [-1.65 to -1.03] | -1.28 [-1.55 to -1.01]
  Phase B, Month 9 | -1.52 [-1.80 to -1.23] | -1.07 [-1.60 to -0.54] | -1.46 [-1.74 to -1.19] | -1.38 [-1.62 to -1.14]
  Phase B, Month 11 | -1.15 [-1.44 to -0.86] | -1.34 [-1.88 to -0.80] | -1.28 [-1.56 to -1.01] | -1.30 [-1.54 to -1.05]
  Phase B, Month 13 | -0.97 [-1.30 to -0.64] | -1.36 [-1.97 to -0.74] | -1.33 [-1.65 to -1.02] | -1.34 [-1.62 to -1.06]
  Phase B, Month 14 | -0.90 [-1.25 to -0.56] | -1.43 [-2.08 to -0.79] | -1.26 [-1.59 to -0.93] | -1.29 [-1.59 to -1.00]

12. Secondary Outcome: Change From Baseline in Sexual Function as Assessed by the SFI: Ejaculation
Description: The SFI is a multidimensional, self-report instrument specifically designed to evaluate sexual function and satisfaction of men on treatment or with conditions that may affect sexual function. It consists of 11 questions which assess patient function in four domains: Sexual drive, Erection, Ejaculation, and Problem assessment, and a question in regards to overall assessment of sexual function.
  Ejaculation domain consist of 2 questions and are scored on a scale of 0-4 (0=minimum, 4=maximum). Total score for the ejaculation domain ranges from 0 to 8. A higher scores represent better sexual function.
Time Frame: During 14 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | DI (Degarelix Intermittent) | DC (Degarelix Continuous) | LC (Leuprolide Continuous) | Total Continuous
Number analyzed (Participants) | 137 | 41 | 150 | 191
Scores on a scale
  Phase A, Month 3 | -1.04 [-1.33 to -0.75] | -0.90 [-1.43 to -0.37] | -0.87 [-1.15 to -0.59] | -0.88 [-1.13 to -0.63]
  Phase A, Month 7 | -1.23 [-1.48 to -0.97] | -0.80 [-1.27 to -0.34] | -1.08 [-1.32 to -0.84] | -1.02 [-1.23 to -0.80]
  Phase B, Month 9 | -1.24 [-1.51 to -0.98] | -1.06 [-1.55 to -0.57] | -0.94 [-1.20 to -0.69] | -0.97 [-1.20 to -0.74]
  Phase B, Month 11 | -0.94 [-1.22 to -0.67] | -1.24 [-1.74 to -0.74] | -0.93 [-1.19 to -0.67] | -1.00 [-1.23 to -0.76]
  Phase B, Month 13 | -0.89 [-1.15 to -0.62] | -1.07 [-1.56 to -0.58] | -1.12 [-1.38 to -0.87] | -1.11 [-1.34 to -0.89]
  Phase B, Month 14 | -0.79 [-1.10 to -0.48] | -1.17 [-1.73 to -0.61] | -0.97 [-1.27 to -0.68] | -1.01 [-1.27 to -0.75]

13. Secondary Outcome: Change From Baseline in Sexual Function as Assessed by the SFI: Problem Assessment
Description: The SFI is a multidimensional, self-report instrument specifically designed to evaluate sexual function and satisfaction of men on treatment or with conditions that may affect sexual function. It consists of 11 questions which assess patient function in four domains: Sexual drive, Erection, Ejaculation, and Problem assessment, and a question in regards to overall assessment of sexual function.
  Problem assessment domain consist of 2 questions and are scored on a scale of 0-4 (0=minimum, 4=maximum). Total score for the problem assessment domain ranges from 0 to 8. A higher scores represent better sexual function.
Time Frame: During 14 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | DI (Degarelix Intermittent) | DC (Degarelix Continuous) | LC (Leuprolide Continuous) | Total Continuous
Number analyzed (Participants) | 137 | 41 | 150 | 191
Scores on a scale
  Phase A, Month 3 | -0.26 [-0.93 to 0.41] | -0.58 [-1.82 to 0.66] | -0.36 [-1.00 to 0.28] | -0.40 [-0.97 to 0.16]
  Phase A, Month 7 | -0.90 [-1.60 to -0.19] | -0.88 [-2.19 to 0.44] | -0.57 [-1.25 to 0.11] | -0.63 [-1.23 to -0.03]
  Phase B, Month 9 | -0.56 [-1.30 to 0.17] | -0.71 [-2.07 to 0.65] | -0.64 [-1.34 to 0.06] | -0.66 [-1.28 to -0.03]
  Phase B, Month 11 | 0.09 [-0.65 to 0.83] | -0.53 [-1.90 to 0.84] | -0.98 [-1.68 to -0.27] | -0.89 [-1.51 to -0.26]
  Phase B, Month 13 | -0.15 [-0.88 to 0.58] | -1.63 [-2.99 to -0.27] | -1.07 [-1.77 to -0.38] | -1.19 [-1.81 to -0.57]
  Phase B, Month 14 | -0.31 [-1.04 to 0.41] | -1.68 [-3.03 to -0.33] | -0.89 [-1.58 to -0.19] | -1.05 [-1.67 to -0.44]

14. Secondary Outcome: Change From Baseline in Sexual Function as Assessed by the SFI: Overall Satisfaction With Sex Life
Description: The SFI is a multidimensional, self-report instrument specifically designed to evaluate sexual function and satisfaction of men on treatment or with conditions that may affect sexual function. It consists of 11 questions which assess patient function in four domains: Sexual drive, Erection, Ejaculation, and Problem assessment, and a question in regards to overall assessment of sexual function.
  Overall satisfaction domain consist of single question and is scored on a scale of 0-4 (0=minimum, 4=maximum). A higher score represent better sexual function.
Time Frame: During 14 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | DI (Degarelix Intermittent) | DC (Degarelix Continuous) | LC (Leuprolide Continuous) | Total Continuous
Number analyzed (Participants) | 137 | 41 | 150 | 191
Scores on a scale
  Phase A, Month 3 | -0.32 [-0.50 to -0.13] | -0.18 [-0.53 to 0.16] | -0.27 [-0.45 to -0.09] | -0.25 [-0.41 to -0.10]
  Phase A, Month 7 | -0.28 [-0.48 to -0.07] | -0.37 [-0.74 to 0.01] | -0.40 [-0.59 to -0.21] | -0.39 [-0.56 to -0.22]
  Phase B, Month 9 | -0.33 [-0.53 to -0.13] | -0.34 [-0.71 to 0.03] | -0.41 [-0.60 to -0.22] | -0.39 [-0.56 to -0.23]
  Phase B, Month 11 | -0.15 [-0.35 to 0.05] | -0.47 [-0.85 to -0.09] | -0.41 [-0.60 to -0.21] | -0.42 [-0.59 to -0.25]
  Phase B, Month 13 | -0.11 [-0.32 to 0.09] | -0.57 [-0.95 to -0.20] | -0.42 [-0.61 to -0.23] | -0.45 [-0.62 to -0.28]
  Phase B, Month 14 | -0.12 [-0.32 to 0.08] | -0.70 [-1.08 to -0.33] | -0.37 [-0.57 to -0.18] | -0.44 [-0.61 to -0.27]

15. Secondary Outcome: Change From Baseline in Sexual Function as Assessed by the SFI: Total SFI Score
Description: The SFI is a multidimensional, self-report instrument specifically designed to evaluate sexual function and satisfaction of men on treatment or with conditions that may affect sexual function. It consists of 11 questions which assess patient function in four domains: Sexual drive, Erection, Ejaculation, and Problem assessment, and a question in regards to overall assessment of sexual function. Total SFI score ranges from 0 to 44. A higher scores represent better sexual function.
Time Frame: During 14 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | DI (Degarelix Intermittent) | DC (Degarelix Continuous) | LC (Leuprolide Continuous) | Total Continuous
Number analyzed (Participants) | 137 | 41 | 150 | 191
Scores on a scale
  Phase A, Month 3 | -4.07 [-5.10 to -3.05] | -3.93 [-5.84 to -2.02] | -3.69 [-4.67 to -2.71] | -3.74 [-4.61 to -2.87]
  Phase A, Month 7 | -5.20 [-6.23 to -4.16] | -4.28 [-6.21 to -2.35] | -4.57 [-5.56 to -3.58] | -4.51 [-5.38 to -3.63]
  Phase B, Month 9 | -4.97 [-6.04 to -3.91] | -4.35 [-6.33 to -2.37] | -4.62 [-5.63 to -3.61] | -4.56 [-5.46 to -3.66]
  Phase B, Month 11 | -3.56 [-4.63 to -2.49] | -4.62 [-6.62 to -2.63] | -4.74 [-5.76 to -3.72] | -4.71 [-5.62 to -3.81]
  Phase B, Month 13 | -3.37 [-4.48 to -2.26] | -5.59 [-7.66 to -3.52] | -5.15 [-6.21 to -4.09] | -5.24 [-6.18 to -4.30]
  Phase B, Month 14 | -3.27 [-4.41 to -2.12] | -5.93 [-8.06 to -3.80] | -4.68 [-5.77 to -3.59] | -4.94 [-5.91 to -3.97]

16. Secondary Outcome: Percentage of Subjects With a Serum PSA Level ≤4.0 ng/mL
Description: Percentage of Subjects With a Serum PSA Level ≤4.0 ng/mL was measured during the study period.
Time Frame: At 14 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | DI (Degarelix Intermittent) | DC (Degarelix Continuous) | LC (Leuprolide Continuous)
Number analyzed (Participants) | 137 | 41 | 150
Percentage of patients | 100 [97.3 to 100] | 97.6 [87.1 to 99.9] | 98.7 [95.3 to 99.8]

17. Secondary Outcome: Time to Return to Testosterone >0.5 ng/mL Level in the DI Treatment Group
Description: The time to testosterone >0.5 ng/mL level in the DI group was counted from the start of Phase B at Day 196 (i.e. 28 days after last injection of degarelix)
Time Frame: During Phase B
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | DI (Degarelix Intermittent)
Number analyzed (Participants) | 137
Days | 112.0 [112.0 to 140.0]

18. Secondary Outcome: Time to Return to Normal Range (≥1.5 ng/mL) or Baseline Testosterone Level
Description: The time to return to normal range (≥1.5 ng/mL) or Baseline testosterone level in the DI group was counted from the start of Phase B at Day 196 (i.e. 28 days after last injection of degarelix).
Time Frame: During Phase B
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | DI (Degarelix Intermittent)
Number analyzed (Participants) | 137
Days | 168 [140.0 to 168.0]

19. Secondary Outcome: Absolute Change From Baseline in Serum Testosterone Levels
Description: Absolute Change From Baseline in Serum Testosterone Levels was measured.
Time Frame: Phase A Visit 1-8 and Phase B Visit 9-15.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | DI (Degarelix Intermittent) | DC (Degarelix Continuous) | LC (Leuprolide Continuous)
Number analyzed (Participants) | 137 | 41 | 150
ng/mL
  Phase A, Visit 1 (Day 0) | NA (NA) — This visit was the first dosing visit. Serum samples were collected pre-dosing on this visit. Thus, the estimated value obtained on this visit were considered as Baseline value. Hence no change is reported. | -2.97 (NA) — One patient erroneously received medication prior to this visit. Thus, the value obtained on this visit was considered as first post-baseline value for this patient and is reported. There was no SD. | NA (NA) — This visit was the first dosing visit. Serum samples were collected pre-dosing on this visit. Thus, the estimated value obtained on this visit were considered as Baseline value. Hence no change is reported.
  Phase A, Visit 2 (Month 1) | -3.64 (1.4) | -3.77 (1.43) | -3.7 (1.56)
  Phase A, Visit 3 (Month 2) | -3.67 (1.4) | -3.77 (1.44) | -3.77 (1.56)
  Phase A, Visit 4 (Month 3) | -3.68 (1.4) | -3.78 (1.43) | -3.77 (1.55)
  Phase A, Visit 5 (Month 4) | -3.67 (1.41) | -3.78 (1.44) | -3.74 (1.61)
  Phase A, Visit 6 (Month 5) | -3.67 (1.41) | -3.78 (1.44) | -3.78 (1.55)
  Phase A, Visit 7 (Month 6) | -3.66 (1.41) | -3.77 (1.44) | -3.77 (1.56)
  Phase A, Visit 8 (Month 7) | -3.66 (1.42) | -3.78 (1.43) | -3.78 (1.55)
  Phase B, Visit 9 (Month 8) | -3.63 (1.44) | -3.76 (1.44) | -3.78 (1.56)
  Phase B, Visit 10 (Month 9) | -3.41 (1.6) | -3.76 (1.44) | -3.78 (1.56)
  Phase B, Visit 11 (Month 10) | -3.0 (1.76) | -3.75 (1.44) | -3.77 (1.57)
  Phase B, Visit 12 (Month 11) | -2.57 (1.78) | -3.74 (1.43) | -3.78 (1.55)
  Phase B, Visit 13 (Month 12) | -2.18 (1.8) | -3.72 (1.43) | -3.78 (1.56)
  Phase B, Visit 14 (Month 13) | -2.1 (1.81) | -3.73 (1.42) | -3.77 (1.57)
  Phase B, Visit 15 (Month 14) | -1.77 (2.27) | -3.71 (1.42) | -3.78 (1.56)

20. Secondary Outcome: Percent Change From Baseline in Serum Testosterone Levels
Description: Percent change from Baseline in serum testosterone levels was measured.
Time Frame: Phase A Visit 1-8 and Phase B Visit 9-15.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | DI (Degarelix Intermittent) | DC (Degarelix Continuous) | LC (Leuprolide Continuous)
Number analyzed (Participants) | 137 | 41 | 150
Percent change
  Phase A, Visit 1 (Day 0) | NA (NA) — This visit was the first dosing visit. Serum samples were collected pre-dosing on this visit. Thus, the estimated value obtained on this visit were considered as Baseline value. Hence no change is reported. | -95.8 (NA) — One patient erroneously received medication prior to this visit. Thus, the value obtained on this visit was considered as first post-baseline value for this patient and is reported. There was no SD. | NA (NA) — This visit was the first dosing visit. Serum samples were collected pre-dosing on this visit. Thus, the estimated value obtained on this visit were considered as Baseline value. Hence no change is reported.
  Phase A, Visit 2 (Month 1) | -96.4 (5.26) | -97.4 (2.31) | -95.5 (4.22)
  Phase A, Visit 3 (Month 2) | -97.3 (2.46) | -97.5 (1.9) | -97.7 (1.44)
  Phase A, Visit 4 (Month 3) | -97.5 (2.06) | -97.8 (1.41) | -97.5 (1.76)
  Phase A, Visit 5 (Month 4) | -97.2 (4.26) | -97.7 (1.58) | -96.2 (14)
  Phase A, Visit 6 (Month 5) | -97.3 (4.42) | -97.6 (2.49) | -97.8 (1.36)
  Phase A, Visit 7 (Month 6) | -96.8 (7.01) | -97.6 (2.03) | -97.9 (1.46)
  Phase A, Visit 8 (Month 7) | -96.9 (6.34) | -97.5 (2.54) | -97.7 (1.67)
  Phase B, Visit 9 (Month 8) | -95.6 (9.69) | -97.1 (3.09) | -97.8 (1.43)
  Phase B, Visit 10 (Month 9) | -88.7 (24.7) | -97 (3.14) | -97.7 (1.7)
  Phase B, Visit 11 (Month 10) | -77 (34.8) | -97 (3.74) | -97.5 (3.49)
  Phase B, Visit 12 (Month 11) | -65.4 (37.7) | -96.7 (3.43) | -97.9 (1.36)
  Phase B, Visit 13 (Month 12) | -54.7 (41.5) | -96 (5.56) | -97.8 (1.45)
  Phase B, Visit 14 (Month 13) | -51.9 (43.1) | -96.5 (3.7) | -97.4 (4.64)
  Phase B, Visit 15 (Month 14) | -44 (66.1) | -95.8 (4.8) | -97.7 (1.56)

ADVERSE EVENTS:
Time Frame: 15 months
Description: Information related to AEs were collected throughout the trial from the time the subject signed the informed consent form till the end of the follow-up period.
Arm/Group | DI (Degarelix Intermittent) | DC (Degarelix Continuous) | LC (Leuprolide Continuous)
Serious Adverse Events (participants affected / at risk) | 26/175 | 6/50 | 18/178
Other Adverse Events (participants affected / at risk) | 159/175 | 47/50 | 158/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | DI (Degarelix Intermittent) (N=175) | DC (Degarelix Continuous) (N=50) | LC (Leuprolide Continuous) (N=178)
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 3
Myocardial infarction (Cardiac disorders) | 2 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 1
Myocardial ischemia (Cardiac disorders) | 1 | 0 | 1
Angina Pectoris (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Peptic ulcer hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 0
Neutropenic infection (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 2
Presyncope (Nervous system disorders) | 2 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1
Dementia (Nervous system disorders) | 0 | 0 | 1
Dementia alzheimer's type (Nervous system disorders) | 1 | 0 | 0
Transient ischemic attack (Nervous system disorders) | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 1
Aortic stenosis (Vascular disorders) | 2 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1
Pelvic venous thrombosis (Vascular disorders) | 1 | 0 | 0
Peripheral ischemia (Vascular disorders) | 0 | 0 | 1
Subclavian steal syndrome (Vascular disorders) | 0 | 0 | 1
Venous insufficiency (Vascular disorders) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0/0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DI (Degarelix Intermittent) (N=175) | DC (Degarelix Continuous) (N=50) | LC (Leuprolide Continuous) (N=178)
Constipation (Gastrointestinal disorders) | 8 (10) | 4 (4) | 12 (12)
Nausea (Gastrointestinal disorders) | 10 (10) | 4 (4) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 9 (10) | 3 (3) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Injection site pain (General disorders) | 79 (284) | 29 (150) | 19 (32)
Fatigue (General disorders) | 30 (41) | 10 (10) | 32 (32)
Injection site erythema (General disorders) | 42 (124) | 17 (56) | 1 (1)
Injection site swelling (General disorders) | 23 (40) | 5 (11) | 0 (0)
Injection site oedema (General disorders) | 6 (15) | 4 (21) | 0 (0)
Pyrexia (General disorders) | 5 (8) | 3 (3) | 2 (2)
Injection site induration (General disorders) | 1 (2) | 3 (16) | 0 (0)
Urinary tract infection (Infections and infestations) | 6 (13) | 4 (7) | 13 (19)
Nasophayrngitis (Infections and infestations) | 7 (9) | 3 (3) | 11 (11)
Upper respiratory tract infection (Infections and infestations) | 7 (8) | 1 (1) | 10 (13)
Sinusitis (Infections and infestations) | 9 (9) | 3 (3) | 3 (3)
Bronchitis (Infections and infestations) | 6 (7) | 3 (3) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 7 (7) | 3 (4) | 10 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (14) | 5 (10) | 17 (27)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 3 (3) | 10 (13)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (18) | 3 (9) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (4) | 3 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 5 (5)
Headache (Nervous system disorders) | 10 (14) | 1 (1) | 9 (10)
Dizziness (Nervous system disorders) | 10 (11) | 2 (2) | 6 (6)
Haematuria (Renal and urinary disorders) | 8 (9) | 4 (4) | 9 (9)
Dysuria (Renal and urinary disorders) | 4 (4) | 3 (3) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (8) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 1 (1)
Hot flush (Vascular disorders) | 87 (91) | 26 (26) | 110 (113)
Hypertension (Vascular disorders) | 12 (12) | 4 (4) | 17 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.